CLINICAL TRIAL: NCT01294059
Title: Effects of Milnacipran on Widespread Mechanical and Thermal Hyperalgesia of Fibromyalgia Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: SAV-MD-06
Record Dates: First submitted 2011-02-09; First posted 2011-02-11 (Estimated); Last update posted 2014-07-31 (Estimated); Status verified 2014-07

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; Hyperalgesia; Pain; Central Sensitization
MeSH Terms: conditions — Fibromyalgia; Hyperalgesia; Pain | interventions — Milnacipran

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sugar pill (Placebo Comparator): One sugar pill twice daily over 6 weeks
  Interventions: Drug: Milnacipran
- Milnacipran (Active Comparator): Milnacipran 50 mg bid over 6 weeks
  Interventions: Drug: Milnacipran

INTERVENTIONS:
Drug: Milnacipran — 50 mg BID Oral x 6 Weeks
  Other Names: Savella

SUMMARY:
Fibromyalgia syndrome (FM) shares many symptoms common to chronic neuropathic pain, including the characteristic hyperalgesia of the skin (thermal, mechanical) and muscles (mechanical) found in almost all FM patients. Milnacipran, a balance norepinephrine-serotonin re-uptake inhibitor, has been found to reduce pain and improve physical function of FM patients. However, little is known about the pain mechanisms that are affected by this medication. Therefore, the investigator wants to determine the efficacy of milnacipran in reducing pain as well as mechanical and thermal hyperalgesia of FM patients during a randomized, double-blind, placebo controlled trial. Because the investigator expects anti-hyperalgesic effects to coincide or precede with effects on clinical FM pain the proposed duration for this trial is 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with diagnosis of chronic wide-spread pain for at least 3 months, who fulfill the 1990 ACR Criteria for FM.
2. Patients with mean pain ratings ≥ 4.0 VAS units, at Screening and Baseline visits.
3. Patients, who are able to comprehend and satisfactorily comply with protocol requirements.
4. Patients who have not taken any pain medications except acetaminophen within 3 days prior to the Baseline Visit (these medications if taken prior to the Screening Visit must be discontinued at Screening Visit and the Baseline Visit may be scheduled at least 7 days past the last dose of these medications).
5. All women of childbearing potential (WOCBP) must have a negative urine pregnancy test at the Screening Visit. All women of childbearing potential participating in the study must use a medically acceptable form of contraception

Exclusion Criteria:

1. FM patients unwilling or unable to discontinue analgesics (except Tylenol) for at least 5 drug half-lives prior to enrollment.
2. Patient has previously failed treatment with Milnacipran for FM pain.
3. Patients who have been treated with MAO inhibitors within 30 days prior to the Baseline Visit.
4. Patients who received ECT within 3 months prior to the Screening Visit.
5. Women who are pregnant or nursing, or women of childbearing potential who do not use adequate contraception, or who are judged to be unreliable in their use of contraception.
6. Patients who have participated in any clinical trial within one month prior to the Screening Visit.
7. Patients who have a medical condition that, in the Investigator's opinion, would expose them to an increased risk of a significant adverse event or interfere with assessments of safety and efficacy during the course of the trial.
8. Patients with severe renal insufficiency (Creatinine clearance < 30 ml/min)
9. Patient has a BDI score >29
10. Patients with any current malignancy, or any clinically significant hematological, endocrine, cardiovascular, renal, hepatic, gastrointestinal or neurological disease (including any form of epilepsy). If there is a history of such disease but the condition has been stable for at least the past year and is judged by the investigator not to interfere with the patient's participation in the study, the patient may be included.
11. Patients with systolic blood pressure greater than 180 mm Hg or less than 90 mm Hg or diastolic blood pressure greater than 105 mm Hg or less than 50 mm Hg at the Screening visit. Similarly, tachycardia of >110/min is exclusionary.
12. Patients who require concomitant therapy with any prohibited prescription or over-the-counter medication, including aspirin (except 81 mg for heart disease) or antidepressant medications.
13. Patients who are unable to speak, read, and understand English or are judged by the investigator to be unable or unlikely to follow the study protocol and complete all scheduled visits.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2009-11; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Mechanical and Heat Hyperalgesia | 2 week intervals

SECONDARY OUTCOMES:
Clinical Pain | daily

CONTACTS AND LOCATIONS:
Overall Officials: Roland Staud, MD, Principal Investigator — University of Florida
Locations (1):
- Center for Musculoskeletal Pain Research, Gainesville, Florida, United States

REFERENCES:
- [Derived] Staud R, Lucas YE, Price DD, Robinson ME. Effects of milnacipran on clinical pain and hyperalgesia of patients with fibromyalgia: results of a 6-week randomized controlled trial. J Pain. 2015 Aug;16(8):750-9. doi: 10.1016/j.jpain.2015.04.010. Epub 2015 May 19. PMID 25998206